CLINICAL TRIAL: NCT03264703
Title: An Observational Study in Patients With Moderated to Severe Rheumatoid Arthritis Who Have Failed to Combination Therapy of Conventional Disease-modifying Antirheumatic Drugs (cDMARDs) to cDMARD Plus Anti-TNF Versus cDMARDs in Real World ["HUMAN" Study]
Brief Title: Study in Patients With Moderated to Severe Rheumatoid Arthritis Who Have Failed to Combination Therapy of Conventional Disease-modifying Antirheumatic Drugs (cDMARDs) to cDMARD Plus ANti-TNF Versus cDMARDs in Real World
Acronym: HUMAN
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: D2E7-M082-601
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Joint pain; Joint stiffness; Joint redness; Loss of joint function; Swollen joints
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with RA with cDMARD, but no anti-TNF experience: Male and female participants diagnosed with rheumatoid arthritis (RA), who have no experience with anti-tumor necrosis factor (anti-TNF) and who have experienced two or more Conventional Disease Modifying Anti-Rheumatic Drugs (cDMARDs) of a stable dose for at least 3 months.

SUMMARY:
This study will be conducted to observe the disease activity change of Conventional Disease Modifying Anti-Rheumatic Drugs (cDMARD) plus anti-tumour necrosis factor (anti-TNF) from baseline to 6 months compared with cDMARDs, as measured by the disease activity score with the erythrocyte sedimentation rate (DAS28-ESR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis within 3 years
* Participants who have no experience with anti-tumor necrosis factor (anti-TNF)
* Participants who have experienced two or more Conventional Disease Modifying Anti-Rheumatic Drugs (cDMARDs) of a stable dose for at least 3 months prior to informed consent
* Participants who change the treatment regimen to one of the following according to the opinion of the investigator:

  1. One cDMARD plus anti-TNF
  2. Two or more cDMARDs: Modifications or additions of cDMARDs that have been treated prior to informed consent

Exclusion Criteria:

* Participants who may be pregnant or lactating women
* Participants who have contraindication to anti-TNF
* Participants who had participated in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female participants diagnosed with rheumatoid arthritis (RA), who have no experience with anti-tumor necrosis factor (anti-TNF) and who have experienced two or more Conventional Disease Modifying Anti-Rheumatic Drugs (cDMARDs) of a stable dose for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the disease activity score 28-erythrocyte sedimentation rate DAS28-ESR at Month 6 | Baseline; Month 6
  DAS28 is a quantitative tool used to measure and monitor disease activity and "the treatment" of rheumatoid arthritis. DAS28 uses a formula that includes the number of tender joints and swollen joints for a maximum of 28 joints. DAS28 is used to assess whether an individual participant has a significant improvement of the disease activity, compared to baseline. A DAS28 score greater than 5.1 implies active disease, a score less than 3.2 implies low disease activity, and a score less than 2.6 implies remission.

SECONDARY OUTCOMES:
Change from Baseline in the DAS28-ESR at Month 3 | Baseline; Month 3
  DAS28 is a quantitative tool used to measure and monitor disease activity and "the treatment" of rheumatoid arthritis. DAS28 uses a formula that includes the number of tender joints and swollen joints for a maximum of 28 joints. DAS28 is used to assess whether an individual participant has a significant improvement of the disease activity, compared to baseline. A DAS28 score greater than 5.1 implies active disease, a score less than 3.2 implies low disease activity, and a score less than 2.6 implies remission.
Change from Baseline in the DAS28-ESR at Month 12 | Baseline; Month 12
  DAS28 is a quantitative tool used to measure and monitor disease activity and "the treatment" of rheumatoid arthritis. DAS28 uses a formula that includes the number of tender joints and swollen joints for a maximum of 28 joints. DAS28 is used to assess whether an individual participant has a significant improvement of the disease activity, compared to baseline. A DAS28 score greater than 5.1 implies active disease, a score less than 3.2 implies low disease activity, and a score less than 2.6 implies remission.
Clinical remission rate measured by DAS28-ESR | Up to 12 months
  Clinical remission is defined as no tender or swollen joints and a normal erythrocyte sedimentation rate. DAS28 will be used to measure disease activity.
Success rates of dose-reduction and discontinuation of steroid(s) | Up to 12 months
  Dose reduction is defined as a reduction by more than 50% compared to baseline.
Scores on the Korean Health Assessment Questionnaire (KHAQ-20), as a measure of quality of life | Up to 12 months
  The KHAQ-20 is a participant-assessed measure of health assessment comprised of 8 indices. Scores for each index range from 0 (no difficulty to do) to 3 (unable to do). The total score is a sum of the 8 index score and ranges from 0 to 24. Higher scores indicate more severe disease.

CONTACTS AND LOCATIONS:
Locations (15):
- South Korea (15):
  - Eisai Trial Site # 1, Ilsan, Gyeonggi-do
  - Eisai Trial Site # 1, Busan
  - Eisai Trial Site # 2, Busan
  - Eisai Trial Site # 3, Busan
  - Eisai Trial Site # 4, Busan
  - Eisai Trial Site # 1, Daegu
  - Eisai Trial Site # 2, Daegu
  - Eisai Trial Site # 1, Seoul
  - Eisai Trial Site # 2, Seoul
  - Eisai Trial Site # 3, Seoul
  - Eisai Trial Site # 4, Seoul
  - Eisai Trial Site # 5, Seoul
  - Eisai Trial Site # 6, Seoul
  - Eisai Trial Site # 7, Seoul
  - Eisai Trial Site # 8, Seoul